CLINICAL TRIAL: NCT01627392
Title: Mechanisms of the Nicotine Metabolism Effect on Tobacco Dependence
Acronym: NMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-08635
Record Dates: First submitted 2012-06-14; First posted 2012-06-25 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smoking abstinence (Experimental)
  Interventions: Behavioral: Smoking abstinence

INTERVENTIONS:
Behavioral: Smoking abstinence — 6 hour smoking abstinence

SUMMARY:
The purpose of the study is to learn more about tobacco dependence and nicotine metabolism in African-Americans and whites, by studying to see if how fast a person metabolizes nicotine (how the body breaks down nicotine into inactive compounds) affects how dependent they are on smoking cigarettes. The investigators believe that people with a faster rate of metabolism may have more severe nicotine withdrawal symptoms and also may have a harder time trying to quit smoking.

DETAILED DESCRIPTION:
Our studies will use the nicotine metabolite ratio (NMR) (the ratio between the nicotine metabolites 3'hydroxycotinine and cotinine)as a simple and clinically feasible biomarker for the rate of nicotine metabolism. The investigators hypothesize that a faster rate of metabolism leads to faster elimination of nicotine from the body and a more rapid dissipation of brain tolerance to nicotine in the interval between cigarettes, leading in turn to (1) more severe nicotine withdrawal symptoms and (2) greater subjective reward from the cigarette smoked following deprivation. These effects would help to explain why smokers with faster rates of nicotine metabolism have a poorer response to smoking cessation therapy when compared to those with slower rates of metabolism.

The investigators will explore the relationship of the NMR to the endophenotypes of withdrawal, craving and reward, with the assumption that these factors are likely intermediaries for the mechanism linking nicotine metabolism to tobacco dependence and smoking cessation rates with pharmacotherapy. Our study design uses a brief (6 hour) interval of smoking abstinence followed by a "reward" cigarette to elicit the subjective responses relating to withdrawal and reward. Because smoking behavior and severity of nicotine dependence vary by race and sex the investigators will also compare the relationship between NMR and withdrawal and reward in African American vs white smokers and in men vs women.

Secondary analyses will examine whether nicotine half-life mediates the observed effects of NMR on primary response measures.

ELIGIBILITY:
Inclusion Criteria:

* African-American or Caucasian
* Age 18-70 years
* Regular smoker of 5 or more cigarettes per day
* Saliva cotinine of 100 ng/ml or greater

Exclusion Criteria:

* Obese (BMI > 38) or underweight (BMI < 17)
* Major systemic or psychiatric condition
* Medications that are inducers of CYP2A6
* History of alcohol abuse
* Positive drug urine tox test
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2012-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Nicotine withdrawal symptoms | 6 hours post nicotine load
  Total withdrawal score as measured by Minnesota Nicotine Withdrawal Scale

SECONDARY OUTCOMES:
Cognitive performance | 6 hours post nicotine load
  Cognitive performance will be measured by n-back computerized testing
Smoking behavior: number of cigarettes | 90 minutes post-abstinence
  Smoking behavior will be measured by number of cigarettes during a monitoring period following the 3rd (reward) cigarette of the protocol
Smoking behavior: number of puffs per cigarette | 90 minutes post-abstinence
  Smoking behavior will be measured by number of puffs per cigarette during a monitoring period following the 3rd (reward) cigarette of the protocol
Smoking behavior: time to first post-reward cigarette | 90 minutes post-abstinence
  Smoking behavior will be measured by time to first post-reward cigarette during a monitoring period following the 3rd (reward) cigarette of the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Neal L Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Nardone N, Shahid M, Strasser AA, Dempsey DA, Benowitz NL. The influence of nicotine metabolic rate on working memory over 6 hours of abstinence from nicotine. Pharmacol Biochem Behav. 2020 Jan;188:172836. doi: 10.1016/j.pbb.2019.172836. Epub 2019 Dec 5. PMID 31812759
- [Derived] Liakoni E, Edwards KC, St Helen G, Nardone N, Dempsey DA, Tyndale RF, Benowitz NL. Effects of Nicotine Metabolic Rate on Withdrawal Symptoms and Response to Cigarette Smoking After Abstinence. Clin Pharmacol Ther. 2019 Mar;105(3):641-651. doi: 10.1002/cpt.1238. Epub 2018 Oct 25. PMID 30242831